CLINICAL TRIAL: NCT03919058
Title: Sit Less or Exercise More: Impact on Cardiometabolic Health in Multiple Sclerosis
Brief Title: Sit Less or Exercise More: Impact on Cardiometabolic Health in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Prof. dr. Bert Op't Eijnde, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RST-MS
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Non-exercise physical activity; NEPA; Cardiometabolic health; Comorbidities
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants will follow four regimes of 4 days each including a control, a sit less, a sit and an exercise regime. The order of the sit and sit less regimes will be randomized. Each activity regime will be followed by a wash-out period of 10 days during which subjects will continue their normal lifestyle.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not know the code of the different regimes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Regime 1: control regime (Active Comparator): All participants start with the control regime, where baseline activity will be measured.
  Interventions: Other: Baseline activity (control regime)
- Regime 2: Sit regime/sit less regime (Experimental): The order of the regimes will be randomized, half of the participants will execute the sit regime as second regime, the other half will execute the sit less regime as second regime. Subjects have to follow a pre-defined activity protocol and receive an activity tracker (Polar M200) in order to self-monitor their activity.
  Interventions: Other: Increased sitting time (sit regime); Other: Non-exercise physical activity (sit less regime)
- Regime 3: Sit less regime/sit regime (Experimental): The order of the regimes will be randomized, half of the participants will execute the sit regime as second regime, the other half will execute the sit less regime as second regime. Subjects have to follow a pre-defined activity protocol and receive an activity tracker (Polar M200) in order to self-monitor their activity.
  Interventions: Other: Increased sitting time (sit regime); Other: Non-exercise physical activity (sit less regime)
- Regime 4: Exercise regime (Experimental): The exercise regime is the final regime for all participants. This is comparable with the sit regime, but 1h of sitting is replaced with 1 exercise bout.
  Interventions: Other: Structured exercise (exercise regime)

INTERVENTIONS:
Other: Baseline activity (control regime) — This is a baseline measurement of physical activity during which subjects will be instructed not to change activity patterns during four days and to note all activities they perform.
  Arms: Regime 1: control regime
Other: Increased sitting time (sit regime) — Participants have to spend 14h of their day sitting, 1h walking and 1h standing, for four consecutive days. According to the compendium of Ainsworth et al. (2011), this corresponds with a daily workload of activities (DWA) of 27 metabolic equivalents (MET's) per day.
  Arms: Regime 2: Sit regime/sit less regime; Regime 3: Sit less regime/sit regime
Other: Non-exercise physical activity (sit less regime) — Each day (4 days in total) will consist of 3h walking, 4h standing and 9h sitting. These time frames are chosen to result in a comparable DWA increase as the exercise regime compared to the sit regime (+7 MET's)27. The additional 2h of walking and 3h of standing, compared to the sitting regime, will be done in a minimum of four bouts with a time interval of > 1h. The subjects will be instructed to walk on a slow pace. i.e. 2-3 km/h (e.g. walking during shopping and work related walking in an office).
  Arms: Regime 2: Sit regime/sit less regime; Regime 3: Sit less regime/sit regime
Other: Structured exercise (exercise regime) — One hour of sitting in the sit regime will be replaced with 1 training session (1h) on a cycle ergometer in the research center. The remaining hours of each day (4 days in total) have to be spent as follows: 13h sitting, 1h walking and 1h standing for daily care. The intensity of the training session (50-60% of Wmax) results in a DWA of 34.5 MET's according to the compendium of physical activities. Duration of training sessions will be adapted individually with ActivPAL data of the sit less and sit regime to identically match DWA increase between the sit less and exercise regime, compared to the sitting regime.
  Arms: Regime 4: Exercise regime

SUMMARY:
This study evaluates the impact of reducing sitting time and increasing exercise time on cardiometabolic health in persons with Multiple Sclerosis.

DETAILED DESCRIPTION:
To date, it is clear that sedentary behaviour is strongly related to an increased risk of type II diabetes, cardiovascular disease and premature mortality. People suffering from chronic disabilities appear to be particularly susceptible to a sedentary lifestyle and inactivity due to primary disease symptoms. To date, this is an important new research topic in Multiple Sclerosis (MS, ~2.3 million people worldwide, ~10-12.000 diagnosed in Belgium) treatment, since previous research reported a significantly higher prevalence of sedentary behaviour in persons with MS (PwMS) compared to healthy controls (HC). PwMS are reported to have a 40% lower daily step count compared to healthy inactive persons and tend to accumulate their sedentary time in longer bouts. As described above and similar to other chronic conditions, a sedentary lifestyle also makes PwMS more vulnerable to the accumulation of important cardiometabolic comorbidities that seem inactivity-related rather than a direct result of non-reversible tissue injury. Such comorbidities include impaired whole body glycaemic control, an abnormal blood lipid profile, an unhealthy body composition and hypertension. In this respect, it is important to note that corticosteroids, which are often used to treat MS patients pharmacologically, elevate fasting glucose and insulin concentrations and induce insulin resistance in HC therefore probably also increase several cardiometabolic risk factors in MS.

Up to now, research in MS has been focused on structured exercise and its positive effects on functional parameters are well-known (e.g. improvements in cardiorespiratory fitness, muscle strength, balance, fatigue, cognition, quality of life and respiratory function). However, evidence is growing that sedentary time, independent of the (dis)practice of structured exercise, is an important independent health risk factor. Consequently, any strategy that also improves cardiometabolic health may help to further optimize rehabilitation in MS. Breaking up and reducing sedentary time with easy, daily activities such as household activities and other activities which increase light-intensity walking and standing, known as non-exercise physical activity (NEPA) may be such a strategy.

NEPA has already been shown to significantly improve cardiometabolic risk markers in healthy, sedentary subjects, type II diabetes patients and obese adults and it involves lower intensity physical activities that are probably more feasible for PwMS. Moreover, with comparable activity workloads, reducing sitting time by NEPA of longer duration decreases insulin levels and fasting lipid levels more than performing one structured exercise bout of moderate intensity that is usually described in current activity guidelines. So far however, acute exercise bouts and NEPA effects on cardiometabolic health in this population have never been described. Therefore, the aim of this study is to investigate whether (1) cardiometabolic health (glycaemic control, blood lipids, inflammation markers and blood pressure) of persons with MS improves when sedentary time is reduced and (2) NEPA results in better cardiometabolic health parameters than (a shorter daily bout of) moderate-intensity exercise when workload of both activities is identical in this population.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men and women ≥18 years old
* Clinical diagnosis of MS (McDonald criteria)
* Expanded Disability Status Score ≤ 5
* Daily internet access

Exclusion Criteria:

* Reported participation in another biomedical trial which may have an effect on blood parameters one month before the pre-study examination or during the study
* Blood donation in the past three months
* Pregnancy or intention of becoming pregnant
* Reported dietary habits: medically prescribed diet, slimming diet
* Reported weight loss (>2kg) in the last three months prior to the screening
* Alcohol use > 20 units per week (during the last 3 months)
* Experimental drug use (during the last 3 months)
* Medication changes (during the last month)
* Medical conditions which make participation in the study not responsible:
* Heart failure: New York Heart Association (NYHA) 3 or higher
* Angina pectoris or signs of cardiac ischemia during exercise testing
* Mental or physical disability
* Based on historical information not able to walk for 3h per day and stand for 4h per day (e.g. intermittent claudication)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Steps per day | Day 1 to 4 of the control regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Day 1 to 4 of the control regime
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Day 1 to 4 of the control regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Day 1 to 4 of the control regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Concentration of glucose | Day after the control regime
  Blood analysis
Concentration of insulin | Day after the control regime
  Blood analysis
Concentration of total cholesterol | Day after the control regime
  Blood analysis
Concentration of high density lipoprotein cholesterol (HDL-cholesterol) | Day after the control regime
  Blood analysis
Concentration of low density lipoprotein cholesterol (LDL-cholesterol) | Day after the control regime
  Blood analysis
Concentration of non-high densitiy lipoprotein cholesterol (non-HDL cholesterol) | Day after the control regime
  Blood analysis
Concentration of triglyceride | Day after the control regime
  Blood analysis
Concentration of apolipoprotein A1 (apo A1) | Day after the control regime
  Blood analysis
Concentration of apolipoprotein B (apo B) | Day after the control regime
  Blood analysis
Concentration of free fatty acids (FFA) | Day after the control regime
  Blood analysis
Concentration of C-reactive protein (CRP) | Day after the control regime
  Blood analysis
Concentration of interleukin 1 (IL-1) | Day after the control regime
  Blood analysis
Concentration of interleukin 6 (IL-6) | Day after the control regime
  Blood analysis
Steps per day | Day 1 to 4 of the Sit regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Dag 1 to 4 of the Sit regime
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Day 1 to 4 of the Sit regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Day 1 to 4 of the Sit regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Concentration of glucose | Day after the Sit regime
  Blood analysis
Concentration of insulin | Day after the Sit regime
  Blood analysis
Concentration of total cholesterol | Day after the Sit regime
  Blood analysis
Concentration of high density lipoprotein cholesterol (HDL-cholesterol) | Day after the Sit regime
  Blood analysis
Concentration of low density lipoprotein cholesterol (LDL-cholesterol) | Day after the Sit regime
  Blood analysis
Concentration of non-high densitiy lipoprotein cholesterol (non-HDL cholesterol) | Day after the Sit regime
  Blood analysis
Concentration of triglyceride | Day after the Sit regime
  Blood analysis
Concentration of apolipoprotein A1 (apo A1) | Day after the Sit regime
  Blood analysis
Concentration of apolipoprotein B (apo B) | Day after the Sit regime
  Blood analysis
Concentration of free fatty acids (FFA) | Day after the Sit regime
  Blood analysis
Concentration of C-reactive protein (CRP) | Day after the Sit regime
  Blood analysis
Concentration of interleukin 1 (IL-1) | Day after the Sit regime
  Blood analysis
Concentration of interleukin 6 (IL-6) | Day after the Sit regime
  Blood analysis
Steps per day | Day 1 to 4 of the Sit Less regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Day 1 to 4 of the Sit Less regime
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Day 1 to 4 of the Sit Less regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Day 1 to 4 of the Sit Less regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Concentration of glucose | Day after the Sit Less regime
  Blood analysis
Concentration of insulin | Day after the Sit Less regime
  Blood analysis
Concentration of total cholesterol | Day after the Sit Less regime
  Blood analysis
Concentration of high density lipoprotein cholesterol (HDL-cholesterol) | Day after the Sit Less regime
  Blood analysis
Concentration of low density lipoprotein cholesterol (LDL-cholesterol) | Day after the Sit Less regime
  Blood analysis
Concentration of non-high densitiy lipoprotein cholesterol (non-HDL cholesterol) | Day after the Sit Less regime
  Blood analysis
Concentration of triglyceride | Day after the Sit Less regime
  Blood analysis
Concentration of apolipoprotein A1 (apo A1) | Day after the Sit Less regime
  Blood analysis
Concentration of apolipoprotein B (apo B) | Day after the Sit Less regime
  Blood analysis
Concentration of free fatty acids (FFA) | Day after the Sit Less regime
  Blood analysis
Concentration of C-reactive protein (CRP) | Day after the Sit Less regime
  Blood analysis
Concentration of interleukin 1 (IL-1) | Day after the Sit Less regime
  Blood analysis
Concentration of interleukin 6 (IL-6) | Day after the Sit Less regime
  Blood analysis
Steps per day | Day 1 to 4 of the Exercise regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Day 1 to 4 of the Exercise regime
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Day 1 to 4 of the Exercise regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Day 1 to 4 of the Exercise regime
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Concentration of glucose | Day after the Exercise regime
  Blood analysis
Concentration of insulin | Day after the Exercise regime
  Blood analysis
Concentration of total cholesterol | Day after the Exercise regime
  Blood analysis
Concentration of high density lipoprotein cholesterol (HDL-cholesterol) | Day after the Exercise regime
  Blood analysis
Concentration of low density lipoprotein cholesterol (LDL-cholesterol) | Day after the Exercise regime
  Blood analysis
Concentration of non-high densitiy lipoprotein cholesterol (non-HDL cholesterol) | Day after the Exercise regime
  Blood analysis
Concentration of triglyceride | Day after the Exercise regime
  Blood analysis
Concentration of apolipoprotein A1 (apo A1) | Day after the Exercise regime
  Blood analysis
Concentration of apolipoprotein B (apo B) | Day after the Exercise regime
  Blood analysis
Concentration of free fatty acids (FFA) | Day after the Exercise regime
  Blood analysis
Concentration of C-reactive protein (CRP) | Day after the Exercise regime
  Blood analysis
Concentration of interleukin 1 (IL-1) | Day after the Exercise regime
  Blood analysis
Concentration of interleukin 6 (IL-6) | Day after the Exercise regime
  Blood analysis

SECONDARY OUTCOMES:
Blood pressure | Day after the Control regime
  Systolic, diastolic and mean arterial blood pressure will be measured 3 times at 5-min intervals using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 2 measurements.
Body weight | Day after the Control regime
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg
Blood pressure | Day after the Sit regime
  Systolic, diastolic and mean arterial blood pressure will be measured 3 times at 5-min intervals using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 2 measurements.
Body weight | Day after the Sit regime
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg
Blood pressure | Day after the Sit Less regime
  Systolic, diastolic and mean arterial blood pressure will be measured 3 times at 5-min intervals using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 2 measurements.
Body weight | Day after the Sit Less regime
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg
Blood pressure | Day after the Exercise regime
  Systolic, diastolic and mean arterial blood pressure will be measured 3 times at 5-min intervals using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 2 measurements.
Body weight | Day after the Exercise regime
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg

CONTACTS AND LOCATIONS:
Overall Officials: Bert Op 't Eijnde, Prof. dr., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

REFERENCES:
- [Derived] Nieste I, Franssen WMA, Duvivier BMFM, Spaas J, Savelberg HHCM, Eijnde BO. Replacing sitting with light-intensity physical activity throughout the day versus 1 bout of vigorous-intensity exercise: similar cardiometabolic health effects in multiple sclerosis. A randomised cross-over study. Disabil Rehabil. 2023 Oct;45(20):3293-3302. doi: 10.1080/09638288.2022.2122601. Epub 2022 Oct 3. PMID 36190113